CLINICAL TRIAL: NCT03286023
Title: Stereotactic Radiotherapy for Patients With Brain Metastases
Brief Title: Stereotactic Radiotherapy for Brain Metastases
Acronym: CKBrainMeta
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Francois Baclesse, Luxembourg (Other)
Responsible Party: Sponsor
Other Study IDs: CYM6 Brain metastases CFB 1
Record Dates: First submitted 2017-09-07; First posted 2017-09-18 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Metastasis Brain
Keywords: brain metastases; stereotactic radiation; cyberknife
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stereotactic radiation: Stereotactic radiation for brain metastases
  Interventions: Radiation: stereotactic radiotherapy

INTERVENTIONS:
Radiation: stereotactic radiotherapy — stereotactic radiotherapy for brain metastases

SUMMARY:
Stereotactic radiotherapy is an innovative treatment enabling to target accurately brain metastases. The aim of this study is to evaluate tumoral response and acute and late toxicity of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Situation 1: in case of several cerebral metastases. In this case, the maximum of cerebral metastases is 3, and the maximum diameter of the largest can not exceed 3 cm. The other two ones can not exceed 1 cm or even maximum 2 cm in diameter for one of the two. The same principle will remain valid in the presence of 2 metastases.
* Situation 2: in the case of a single metastasis, the diameter should be a maximum of 3 cm
* Situation 3: in case of metastasis supposed to be radioresistant (renal adenocarcinoma, sarcoma, melanoma ...), only a single metastasis of not more than 3 cm in diameter will be accepted. A primary resection followed by radiotherapy will be preferred.
* Situation 4: In case of localization near a structure at risk (contact with anterior optical pathways, central nuclei or the brainstem or localization in these structures), a maximum number of 3 metastases may be accepted. However, that included in or close to the risk structure can not exceed 2 cm in diameter and the other two, located outside a risk structure will have a diameter not exceeding 1 or even maximum 2 cm.
* Situation 5: single metastasis of maximum 3 cm in a context of re-irradiation, the whole encephalon having already received the dose of 10 X 3 Gy or its biological equivalent of dose.
* Signed informed consent

Exclusion Criteria:

* Impossibility of performing an MRI or a CT-scan of the brain with injection of contrast agent
* Metastases greater than 3 cm at the start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain metastases
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-10; Primary Completion 2019-10 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tumoral response | 4 weeks after treatment
  Evaluation of response using Magnetic resonance imaging (Recist criteria)
Evaluation of tumoral response | 8 weeks after treatment
  Evaluation of response using Magnetic resonance imaging (Recist criteria)

SECONDARY OUTCOMES:
Evaluation of toxicity | 1, 3, 6, 9, 12, 15 months after treatment
  Evaluation of toxicity using CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Francois Baclesse, Esch-sur-Alzette, SUD, Luxembourg

IPD SHARING:
Plan to Share IPD: No